CLINICAL TRIAL: NCT05563688
Title: Effect of Acute Sleep Restriction on Responses to Hypoxia
Acronym: HypSom
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PBMD09; 2022-A00464-39 (Other: IDRCB)
Record Dates: First submitted 2022-09-16; First posted 2022-10-03 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Sleep Deprivation; Hypoxia
MeSH Terms: conditions — Sleep Deprivation; Hypoxia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hypoxia exposure — Each participant will be exposed to the hypoxic environment on 2 occasions (one after a normal sleep night and one after sleep deprivation).
  Each exposure will be for 5 hours at a FiO2 of 13.2% (3500 m simulated altitude).
  This exposure will be carried out in a normobaric hypoxic tent (Sporting Edge®).
Other: Sleep deprivation — Each participant will be exposed to sleep deprivation on 2 occasions (one before normoxia exposure and one before hypoxia exposure).
  Each sleep deprivation involves a time spent in bed of 3 hours (03h00 - 06h00). Sleep deprivation will be carried out in a sleep apartment. Sleep duration and quality will be assessed using a sleep headband (Dreem®), actigraphs Actiwatch® and E4 Empatica®) and a sleep diary.
Behavioral: Cognitive tasks — Participants will perform several cognitive tasks in the following conditions:
  * in normoxia (FiO2 = 21%) after a night of usual sleep (> 6 hours) ;
  * in normoxia (FiO2 = 21%) after a night of reduced sleep (3 hours);
  * in normobaric hypoxia (FiO2 = 13.2%) after a night of normal sleep (> 6 hours);
  * in normobaric hypoxia (FiO2 = 13.2%) after a night of reduced sleep (3 hours).

SUMMARY:
At altitude, humans are exposed to environmental hypoxia induced by the decrease in barometric pressure. On duty or in training, mountain troops, paratroopers or aircrew are regularly exposed to altitude. The effects of altitude on humans occur gradually from 1500 m and depend on both the duration of exposure and the altitude level. Cognitive disorders can occur from 3500 m (threshold of disorders) but there is a very large inter-individual variability.

The countermeasure to altitude hypoxia is oxygen but its use is not systematic between 3000 and 4000 m. Its use depends on the duration of exposure, without clearly established standards. Incapacitating effects on the operational capacity and health of soldiers can therefore occur as early as 3500 m.

In operations or during training, altitude exposure is often associated with a significant sleep debt (particularly during night or early morning missions), jet lag or precarious rest conditions in overseas operations. These sleep restrictions promote the degradation of mental performance with effects similar to those observed in hypoxia.

The combination of these constraints induces a physiological stress which can favour alterations in mental performance, an increase in incapacity, intolerance to altitude or the occurrence of altitude-related pathologies in military personnel. This could occur in particular in the operational zone around the threshold of disorders (3500 m) where the indication of oxygen is discussed.

The objective of this study is to assess the impact of acute sleep restriction on hypoxia tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Healthy
* Between 18 and 45
* Smoking < 5 cigarettes per day or nicotine-free electronic cigarette
* Having regular physical activity (between 1 and 4 hours of physical activity per week)
* Affiliated or entitled to a social security plan
* No contraindication to physical exercise
* Having given their consent

Exclusion Criteria:

* Female
* BMI > 30
* Active medical pathology (cardiological, renal, hepatic, cutaneous, neurological, etc.),
* History of active pathology of less than 6 months
* Significant deviation with the normal values observed during the interrogation, clinical examination or electrocardiogram
* Having spent time at altitude (> 3500 m) during the last 3 months
* Absolute or relative contraindication to a stay at high altitude
* Medical contraindication to sport practice
* Skin allergy to modified ethanol or capsaicin
* Wearing a pacemaker or ferromagnetic implants
* Poor venous capital
* Pittsburgh Sleep Quality Index Questionnaire > 5
* Usual sleep duration < 6 hours
* Not covered by a health insurance plan

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be composed of healthy active young men.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Mean reaction time (in ms) to the 10-minute psychomotor vigilance task (PVT-10), at the end of the exposure. | Through study completion (20.5 months)
  PVT-10 is a sustained-attention, reaction-timed task that measures the consistency with which subjects respond to a visual stimulus.
  The participant sits in front of a computer. He has a screen in front of him with a 4-digit counter (0 at the start). He is instructed to click the left mouse button as fast as possible when the counter starts to scroll. The counter returns to zero when the participant has clicked.
  Reaction time (in ms) is calculated for each stimulus.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pontiggia A, Quiquempoix M, Fabries P, Beauchamps V, Jacques C, Guillard M, Van Beers P, Malle C, Gomez-Merino D, Koulmann N, Chennaoui M, Sauvet F; HYPSOM Investigator Group. Robust multimodal mental workload classification: A cross-physiological condition machine learning approach. Comput Methods Programs Biomed. 2026 Jan 14;277:109251. doi: 10.1016/j.cmpb.2026.109251. Online ahead of print. PMID 41576780